CLINICAL TRIAL: NCT03486990
Title: A Phase 1, First-in-Human, 2-Part, Multicenter Dose Escalation and Repeat Dose Study of the Safety, Tolerability and Pharmacokinetics of TIMP-GLIA in Subjects With Celiac Disease
Brief Title: Study of the Safety, Tolerability and Pharmacokinetics of TIMP-GLIA in Subjects With Celiac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: COUR Pharmaceutical Development Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TGLIA-5.001
Record Dates: First submitted 2018-03-21; First posted 2018-04-03 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Celiac Disease
Keywords: safety; tolerability; pharmacokinetics; celiac; gliadin; gluten
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: Single ascending dose followed by repeat dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A, Cohort 1: 0.1 mg/kg (Experimental): TIMP-GLIA 0.1 mg/kg, infusion, intravenously, once on Day 1.
  Interventions: Drug: TIMP-GLIA
- Part A, Cohort 2: 0.5 mg/kg (Experimental): TIMP-GLIA 0.5 mg/kg, infusion, intravenously, once on Day 1.
  Interventions: Drug: TIMP-GLIA
- Part A, Cohort 3: 1.0 mg/kg (Experimental): TIMP-GLIA 1.0 mg/kg, infusion, intravenously, once on Day 1.
  Interventions: Drug: TIMP-GLIA
- Part A, Cohort 4: 2.0 mg/kg (Experimental): TIMP-GLIA 2.0 mg/kg, infusion, intravenously, once on Day 1.
  Interventions: Drug: TIMP-GLIA
- Part A, Cohort 5: 4.0 mg/kg (Experimental): TIMP-GLIA 4.0 mg/kg, infusion, intravenously, once on Day 1.
  Interventions: Drug: TIMP-GLIA
- Part A, Cohort 6: 8.0 mg/kg (Experimental): TIMP-GLIA 8.0 mg/kg, infusion, intravenously, once on Day 1.
  Interventions: Drug: TIMP-GLIA
- Part B, Cohort 1: 2.0 mg/kg (Experimental): TIMP-GLIA 2.0 mg/kg, infusion, intravenously, once on Days 1 and 8.
  Interventions: Drug: TIMP-GLIA
- Part B, Cohort 2: 4.0 mg/kg (Experimental): TIMP-GLIA 4.0 mg/kg, infusion, intravenously, once on Days 1 and 8.
  Interventions: Drug: TIMP-GLIA
- Part B, Cohort 3: 8.0 mg/kg (Experimental): TIMP-GLIA 8.0 mg/kg, infusion, intravenously, once on Days 1 and 8.
  Interventions: Drug: TIMP-GLIA

INTERVENTIONS:
Drug: TIMP-GLIA — intravenous infusion.
  Other Names: TAK-101

SUMMARY:
This study is to characterize the safety and tolerability of an investigational drug called TIMP-GLIA when either one or two intravenous doses are given to subjects with celiac disease. The way the body reacts to TIMP-GLIA is being checked by laboratory tests of the blood and urine, and study subject health will also be monitored by vital signs such as blood pressure, electrocardiogram (ECG), and physical examination.

DETAILED DESCRIPTION:
This study is a 2-part, multicenter study. In Part A, eligible subjects will be enrolled into escalating dose cohorts (n = 2/cohort for 2 dose levels followed by n = 3/cohort for 4 dose levels). TIMP-GLIA will be administered as a single intravenous (IV) infusion on Day 1. A staggered dosing strategy will be used in Part A. Subjects will undergo medical observation in the clinic for at least 48 hours after dosing and participate in outpatient follow-up visits. Adverse events (AEs), vital signs, and electrocardiograms (ECGs) and laboratory data (serum chemistry, coagulation, hematology and urinalysis, cytokines) will be assessed by a Safety Committee before the next cohort will be dosed at a higher dose level.

After completion of Part A and confirmation by the Safety Committee to proceed, eligible subjects (n=3) will receive two IV infusions of TIMP-GLIA, 7 days apart, on Day 1 and on Day 8. Each subject in Part B will be observed in clinic for 48 hours after each dose and undergo similar testing and follow-up visits as in Part A.

The safety and pharmacokinetic profile of TIMP-GLIA will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* The subject provides written informed consent and is willing and able to comply with study requirements.
* At screening the subject has a minimum body mass index (BMI) of 16 kg/m2 and a minimum body weight of 33 kg up to a maximum body weight of 129 kg, inclusive. If subject is considered to be underweight or overweight/obese, the subject is otherwise healthy in the opinion of the investigator.
* The subject has celiac disease characterized at Screening Visit by:
* a history of biopsy-confirmed celiac disease; and
* no known gluten exposure for at least 10 days; and
* willingness to maintain a gluten-free diet for the duration of the study; and
* a negative or weak positive transglutaminase (tTG)-specific IgA titer if the subject has a normal total immunoglobulin A (IgA) titer or has a partial IgA deficiency OR
* a negative or weak positive deamidated gliadin peptide (DGP)-specific immunoglobulin G (IgG) titer if the subject has IgA deficiency.
* The male subject or female subject of childbearing potential will practice medically approved contraception during the study.

Exclusion Criteria:

* The subject has a history of clinically confirmed immunoglobulin E-mediated reaction and/or anaphylaxis to wheat (i.e., "wheat allergy"), barley or rye.
* The subject has a known history of hypersensitivity or allergies to TIMP-GLIA components OR any other known severe hypersensitivity or allergic reaction (resulted in hospitalization [initial or prolonged], congenital anomaly, or disability, or that required medical intervention to prevent permanent impairment or damage) to any other allergens (medications, food or environmental).
* The subject has uncontrolled celiac disease and/or complications of celiac disease, or otherwise has experienced celiac symptomology within 10 days of screening, in the opinion of the investigator.
* The subject has a history of, or has an active, significant, clinically relevant, comorbidity (including Type 1 and Type 2 diabetes mellitus and other autoimmune disorders, splenectomy) that, in the opinion of the investigator, would make the subject unsuitable for participation in the study and/or could adversely affect interpretation of the study results.
* The subject has had significant changes to or anticipates changes to prescription or non-prescription medication used to manage an underlying comorbidity within 30 days prior to first dosing (Day 1).
* The subject is currently taking or received systemic biologics 6 months prior to first dosing (Day 1).
* The subject has a compromised immune system, e.g.
* known human immunodeficiency virus (HIV) infection or positive for HIV antibodies at Screening or
* immunosuppressive medical treatment taken during the 2 months prior to first dosing (Day 1) or
* immunosuppressive doses of corticosteroids (more than 20 mg of prednisone given daily for 2 weeks or more within 2 months prior to first dosing (Day 1), or any dose of corticosteroids within 30 days of first dosing (Day 1), or high dose inhaled corticosteroids [>960 µg/day of beclomethasone dipropionate or equivalent]) within 30 days of first dosing Day 1.
* The subject has currently untreated or active gastrointestinal disease such as peptic ulcer disease, esophagitis (Los Angeles Classification ≥ Grade C), irritable bowel syndrome, inflammatory bowel disease, or microscopic colitis.
* The subject has an active malignancy, or history of malignancy or chemotherapy, within the past 5 years other than history of localized or surgical removal of focal basal cell skin cancer, cervical cancer in situ treated successfully in the past by local treatment (including but not limited to cryotherapy or laser therapy) or by hysterectomy.
* The subject has known liver disease or serology positive for hepatitis C infection; positive hepatitis B surface antigen (HBsAg) at Screening Visit.
* The subject has a positive test result for drugs of abuse, cannabinoids, or alcohol at Screening Visit or at Check-in.
* The subject has a history of any drug or alcohol abuse in the past 5 years or alcohol consumption habits that, in the opinion of the investigator, would interfere with the subject's ability to comply with the study requirements.
* The subject has clinically significant laboratory test results (e.g., liver tests) or electrocardiogram (EGC) abnormalities (e.g., cardiac conduction abnormalities) at Screening
* The subject received a live or inactive vaccine within 28 days prior or a subunit vaccine within 14 days prior to first dosing/Day 1 or the subject has a planned vaccination during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (4):
- United States (4):
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Mass General Hospital Translational and Clinical Research Centers, Boston, Massachusetts
  - Mayo Gastroenterology Research Unit, Rochester, Minnesota
  - Prism Clinical Research, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Kelly CP, Murray JA, Leffler DA, Getts DR, Bledsoe AC, Smithson G, First MR, Morris A, Boyne M, Elhofy A, Wu TT, Podojil JR, Miller SD; TAK-101 Study Group. TAK-101 Nanoparticles Induce Gluten-Specific Tolerance in Celiac Disease: A Randomized, Double-Blind, Placebo-Controlled Study. Gastroenterology. 2021 Jul;161(1):66-80.e8. doi: 10.1053/j.gastro.2021.03.014. Epub 2021 Mar 17. PMID 33722583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 23 January 2018 to 22 July 2019.
Pre-assignment Details: Participants diagnosed with celiac disease (CD) were enrolled to receive TIMP-GLIA as a single dose escalation of 0.1 milligram per kilogram (mg/kg), 0.5 mg/kg, 1.0 mg/kg, 2.0 mg/kg, 4.0 mg/kg, 8.0 mg/kg in Part A; and TIMP-GLIA as a two dose escalation of 2.0 mg/kg, 4.0 mg/kg, 8.0 mg/kg in Part B.
Period: Overall Study
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Started | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Completed | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population, included all participants who signed the study-specific informed consent document and received at least 1 dose of TIMP-GLIA.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg | Total
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (27.58) | 53.5 (20.51) | 39.3 (15.57) | 38.0 (4.58) | 48.3 (14.19) | 27.5 (4.65) | 42.5 (13.44) | 53.5 (7.78) | 32.5 (2.12) | 40.3 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 3 | 3 | 2 | 2 | 1 | 18
  Male | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Day 180
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Participants
  TEAEs | 1 | 2 | 3 | 3 | 2 | 3 | 1 | 1 | 2
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Grade 3 or Higher TEAEs and Drug-related Adverse Events
Description: AE Grades will be evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE), version 4.0. Grade 1 scaled as Mild; Grade 2 scaled as Moderate; Grade 3 scaled as severe or medically significant but not immediately life-threatening; Grade 4 scaled as life-threatening consequences; and Grade 5 scaled as death related to AE. Drug-related adverse events are those that the investigator assessed as possibly or probably related to the study treatment.
Time Frame: From Day 1 up to Day 180
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Participants
  Grade 3 or Higher TEAEs | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Drug-related Adverse Events | 1 | 0 | 2 | 2 | 2 | 3 | 0 | 1 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Time Frame: From Day 1 up to Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Electrocardiograms (ECG) Findings
Time Frame: From Day 1 up to Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Arterial Oxygen Saturation Levels
Time Frame: From Day 1 up to Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs Values
Time Frame: From Day 1 up to Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C1q Binding at Day 3
Description: Baseline is defined as Day 1 pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and Day 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units per milliliter (U/ml)
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
units per milliliter (U/ml)
  Baseline (Day 1 pre-dose) | 2.15 (0.495) | 2.85 (0.778) | 3.30 (0.990)
  Change at Day 3 | 1.20 (0.000) | 0.60 (0.141) | -0.35 (0.071)

8. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C1q Binding at Day 7
Description: Baseline is defined as Day 1 pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and Day 7
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
U/ml
  Baseline (Day 1 pre-dose) | 2.15 (0.495) | 2.85 (0.778) | 3.30 (0.990)
  Change at Day 7 | 0.75 (0.071) | 0.00 (0.000) | 0.85 (1.344)

9. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C1q Binding at Day 8
Description: Baseline is defined as Day 1 pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and Day 8
Population: The safety population, included all participants who signed the study-specific informed consent document and received at least 1 dose of TIMP-GLIA. The safety analysis population where data at specified time points were available.
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
U/ml
  Baseline (Day 1 pre-dose) | 2.15 (0.495) | 2.85 (0.778) | 3.30 (0.990)
  Change at Day 8: number analyzed (Participants) | 2 | 1 | 2
  Change at Day 8 | 0.70 (0.141) | 0.10 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 1.50 (1.838)

10. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C1q Binding at Day 10
Description: Baseline is defined as Day 1 pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and Day 10
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
U/ml
  Baseline (Day 1 pre-dose) | 2.15 (0.495) | 2.85 (0.778) | 3.30 (0.990)
  Change at Day 10 | 1.85 (0.778) | 1.00 (1.273) | 1.25 (1.485)

11. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C1q Binding at Day 14
Description: Baseline is defined as Day 1 pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and Day 14
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
U/ml
  Baseline (Day 1 pre-dose) | 2.15 (0.495) | 2.85 (0.778) | 3.30 (0.990)
  Change at Day 14 | 0.90 (0.141) | 1.65 (0.495) | 1.30 (1.273)

12. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C1q Binding at Day 38
Description: Baseline is defined as Day 1 pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and Day 38
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
U/ml
  Baseline (Day 1 pre-dose) | 2.15 (0.495) | 2.85 (0.778) | 3.30 (0.990)
  Change at Day 38: number analyzed (Participants) | 1 | 2 | 2
  Change at Day 38 | 0.30 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 1.50 (1.273) | 1.00 (1.980)

13. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C1q Binding at Day 60
Description: Baseline is defined as Day 1 pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and Day 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
U/ml
  Baseline (Day 1 pre-dose) | 2.15 (0.495) | 2.85 (0.778) | 3.30 (0.990)
  Change at Day 60 | 0.65 (0.354) | 1.15 (1.061) | 1.10 (1.838)

14. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C3a and SC5B-9 Levels at 15 Minutes Post-dose on Day 1
Description: Baseline was defined as Day 1 Pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and 15 minutes (min) post-dose on Day 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
nanogram per milliliter (ng/mL)
  Baseline (Day 1 pre-dose): C3a level | 32.25 (23.264) | 16.15 (0.636) | 18.65 (17.041)
  Change at 15 min post-dose on Day 1: C3a level | 45.40 (43.841) | 134.90 (104.369) | 46.25 (13.930)
  Baseline (Day 1 pre-dose): SC5B-9 level | 109.5 (17.68) | 95.5 (33.23) | 112.0 (33.94)
  Change at 15 min post-dose on Day 1: SC5B-9 level | 59.0 (49.50) | 196.0 (193.75) | 130.5 (33.23)

15. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C3a and SC5B-9 Levels at 30 Minutes Post-dose on Day 1
Description: Baseline was defined as Day 1 Pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and 30 min post-dose on Day 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
ng/mL
  Baseline (Day 1 pre-dose): C3a level | 32.25 (23.264) | 16.15 (0.636) | 18.65 (17.041)
  Change at 30 min post-dose on Day 1: C3a level | 87.50 (56.569) | 144.00 (11.455) | 65.65 (34.719)
  Baseline (Day 1 pre-dose): SC5B-9 level | 109.5 (17.68) | 95.5 (33.23) | 112.0 (33.94)
  Change at 30 min post-dose on Day 1: SC5B-9 level | 179.0 (2.83) | 307.0 (41.01) | 293.0 (185.26)

16. Primary Outcome: Part B: Change From Baseline (Day 1 Pre-dose) in C3a and SC5B-9 Levels at Day 2
Description: Baseline was defined as Day 1 Pre-dose.
Time Frame: Baseline (Day 1 pre-dose) and Day 2
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 2
ng/mL
  Baseline (Day 1 pre-dose): C3a level | 32.25 (23.264) | 16.15 (0.636) | 18.65 (17.041)
  Change at Day 2: C3a level | -6.55 (12.092) | 0.90 (0.990) | -6.70 (20.789)
  Baseline (Day 1 pre-dose): SC5B-9 level | 109.5 (17.68) | 95.5 (33.23) | 112.0 (33.94)
  Change at Day 2: SC5B-9 level | 26.0 (14.14) | -12.5 (36.06) | 2.0 (22.63)

17. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Hematology, Serum Chemistry, Coagulation, and Urinalysis
Time Frame: From Day 1 up to Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Part A (Greater Than or Equal to [>=] 4.0 mg/kg) and Part B: Number of Participants With Clinically Significant Change From Baseline in Gliadin-Specific T-cell Proliferation and Cytokine Release Markers
Time Frame: Part A (>=4.0 mg/kg): Day 1 pre-dose up to 144 hours post-dose on Day 7; Part B: Day 8 pre-dose up to 144 hours post-dose on Day 14
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 3 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Time Frame: From Day 1 up to Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

20. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration For TIMP-GLIA
Time Frame: Parts A and B, Day 1: pre-dose and at multiple time points (up to 144 hours) post-dose; Part B, Day 8: pre-dose and at multiple time points (up to 144 hours) post-dose
Population: The pharmacokinetic (PK) population who received at least 1 dose of TIMP-GLIA and had at least 1 PK parameter reported. The PK analysis population where data at specified time points were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2
nanogram per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 2 | 3 | 3 | 3 | 0 | 2 | 2 | 2
  Day 1 | 91.8 (48.4) | 220 (3.0) | 457 (17.6) | 845 (23.6) |  | 252 (6.7) | 529 (22.6) | 938 (2.9)
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Day 8 |  |  |  |  |  | NA (NA) — Data was not calculated in more than 1/3 of participants due to poor or incomplete profile and not estimable in WinNonLin, or Percent of area under the plasma concentration-time curve extrapolated to infinity (%AUCextrap) exceeds 25%. | 408 (26.8) | 735 (11.7)

21. Secondary Outcome: Clast: Last Measurable Observed Plasma Concentration For TIMP-GLIA
Time Frame: as for outcome 20
Population: The PK population who received at least 1 dose of TIMP-GLIA and had at least 1 PK parameter reported. The PK analysis population where data at specified time points were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2
ng/mL
  Day 1 | 50.6 (12.2) | 63.9 (29.2) | 68.6 (27.2) | 55.8 (30.2) | 77.2 (23.7) | 97.9 (85.1) | 47.9 (19.0) | 111 (5.7)
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Day 8 |  |  |  |  |  | NA (NA) — Data was not calculated in more than 1/3 of participants due to poor or incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 133 (137.7) | 54.4 (19.5)

22. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TIMP-GLIA
Time Frame: as for outcome 20
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2
hour
  Day 1: number analyzed (Participants) | 2 | 3 | 3 | 3 | 0 | 2 | 2 | 2
  Day 1 | 0.54 [0.50 to 0.58] | 0.50 [0.50 to 0.58] | 0.50 [0.50 to 0.58] | 0.50 [0.50 to 0.58] |  | 2.86 [2.85 to 2.87] | 3.21 [2.82 to 3.60] | 2.94 [2.83 to 3.05]
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Day 8 |  |  |  |  |  | NA [NA to NA] — Data was not calculated in more than 1/3 of participants due to poor or incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 3.08 [2.82 to 3.33] | 2.90 [2.80 to 3.00]

23. Secondary Outcome: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TIMP-GLIA
Time Frame: as for outcome 20
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2
hour*nanogram per milliliter (h*ng/mL)
  Day 1: number analyzed (Participants) | 0 | 2 | 2 | 3 | 2 | 1 | 2 | 2
  Day 1 |  | 604 (3.4) | 3100 (27.0) | 3170 (22.8) | 8430 (48.9) | NA (NA) — Data was not calculated in more than 1/3 of participants due to poor or incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 3220 (31.5) | 5080 (9.2)
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Day 8 |  |  |  |  |  |  | NA (NA) — Data was not calculated in more than 1/3 of participants due to poor or incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 3250 (15.1)

24. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TIMP-GLIA
Time Frame: as for outcome 20
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2
h*ng/mL
  Day 1 | 119 (210.7) | 503 (12.1) | 1690 (88.1) | 2920 (21.6) | 2870 (501.3) | 932 (65.2) | 2930 (30.6) | 4590 (9.6)
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Day 8 |  |  |  |  |  | NA (NA) — Data was not calculated in more than 1/3 of participants due to poor or incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 1410 (107.1) | 3050 (14.7)

25. Secondary Outcome: Tlast: Time to Reach the Last Measurable Plasma Concentration for TIMP-GLIA
Time Frame: as for outcome 20
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2
hour
  Day 1 | 2.49 [1.00 to 3.98] | 4.00 [4.00 to 4.00] | 12.17 [4.00 to 24.00] | 12.00 [12.00 to 12.17] | 12.00 [4.02 to 24.53] | 7.99 [4.00 to 11.98] | 18.10 [12.20 to 24.00] | 12.00 [12.00 to 12.00]
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Day 8 |  |  |  |  |  | NA [NA to NA] — Data was not calculated in more than 1/3 of participants due to poor or incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 8.01 [4.02 to 12.00] | 12.08 [12.00 to 12.15]

26. Secondary Outcome: T1/2: Terminal Phase Elimination Half-life (T1/2) for TIMP-GLIA
Time Frame: as for outcome 20
Population: as for outcome 21
Measure: Median (Full Range); unit: hour
Arm/Group | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2
hour
  Day 1: number analyzed (Participants) | 1 | 3 | 3 | 3 | 2 | 1 | 2 | 2
  Day 1 | NA [NA to NA] — Data was not calculated in more than 1/3 of participants due to poor or incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 1.81 [1.63 to 2.57] | 4.38 [1.92 to 8.24] | 3.03 [2.86 to 3.35] | 4.36 [2.72 to 6.00] | NA [NA to NA] — Parameter was not estimable in more than 1/3 of participants due to poor/incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 4.60 [2.77 to 6.43] | 3.03 [3.02 to 3.04]
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Day 8 |  |  |  |  |  |  | NA [NA to NA] — Parameter was not estimable in more than 1/3 of participants due to poor/incomplete profile and not estimable in WinNonLin, or %AUCextrap exceeds 25%. | 2.51 [2.46 to 2.56]

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of study drug up to Day 180
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part A, Cohort 1: 0.1 mg/kg | Part A, Cohort 2: 0.5 mg/kg | Part A, Cohort 3: 1.0 mg/kg | Part A, Cohort 4: 2.0 mg/kg | Part A, Cohort 5: 4.0 mg/kg | Part A, Cohort 6: 8.0 mg/kg | Part B, Cohort 1: 2.0 mg/kg | Part B, Cohort 2: 4.0 mg/kg | Part B, Cohort 3: 8.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/3 | 0/3 | 0/3 | 0/4 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3 | 0/3 | 0/3 | 0/4 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 3/3 | 3/3 | 2/3 | 3/4 | 1/2 | 1/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Cohort 1: 0.1 mg/kg (N=2) | Part A, Cohort 2: 0.5 mg/kg (N=2) | Part A, Cohort 3: 1.0 mg/kg (N=3) | Part A, Cohort 4: 2.0 mg/kg (N=3) | Part A, Cohort 5: 4.0 mg/kg (N=3) | Part A, Cohort 6: 8.0 mg/kg (N=4) | Part B, Cohort 1: 2.0 mg/kg (N=2) | Part B, Cohort 2: 4.0 mg/kg (N=2) | Part B, Cohort 3: 8.0 mg/kg (N=2)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue geographic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gluten sensitivity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT03486990/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT03486990/SAP_001.pdf